CLINICAL TRIAL: NCT02282735
Title: Parental Decision-Making for Children With Relapsed Neuroblastoma
Status: Active, not recruiting | Type: Observational
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Jennifer Mack, MD, Attending Physician, Pediatric Oncology, Dana-Farber Cancer Institute
Other Study IDs: 13-083
Record Dates: First submitted 2014-10-30; First posted 2014-11-04 (Estimated); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Relapsed Neuroblastoma
Keywords: neuroblastoma; end-of-life; decision-making; parent; child; prognosis; preferences; childhood cancer; oncology
MeSH Terms: conditions — Neuroblastoma; Death; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Parental decision-making for children with advanced cancer is complex. Many parents have overly optimistic beliefs about prognosis and as a result choose aggressive measures even at the end of life, which are associated with greater suffering. Yet most parents wish to limit suffering, and in retrospect, many regret choices for cancer treatment for advanced cancer. These findings suggest that parents do not always have the information they need to make decisions that reflect their preferences.

The proposed study will evaluate parental decision-making in advanced cancer, addressing gaps in the literature in 3 important respects. 1) Previous work on decision-making for children with advanced cancer has typically looked at decisions at one point in time, often asking parents to reflect on decisions after the child's death, even though parents' understanding of prognosis and decisions about care evolve over time. We will evaluate parental decision-making for advanced cancer over time. 2) Existing work focuses on aggressive end-of-life care as the worst possible outcome. However, some parents wish to pursue aggressive measures even when they recognize that the child has little chance for cure. We will evaluate the extent to which parental decision-making is informed and consonant with preferences, regardless of whether decisions lead to aggressive or palliative care. 3) Previous studies have focused on groups of different childhood cancers, making it difficult to ascertain whether differences in decision-making reflect differences in diseases, options for care, or parent preferences. We will focus on a single disease, relapsed neuroblastoma, as a model for parental decision-making.

DETAILED DESCRIPTION:
Parental decision-making for children with advanced cancer is complex. Many parents have overly optimistic beliefs about prognosis and as a result choose aggressive measures even at the end of life, which are associated with greater suffering. Yet most parents wish to limit suffering, and in retrospect, many regret choices for cancer treatment for advanced cancer. These findings suggest that parents do not always have the information they need to make decisions that reflect their preferences.

The proposed study will evaluate parental decision-making in advanced cancer, addressing gaps in the literature in 3 important respects. 1) Previous work on decision-making for children with advanced cancer has typically looked at decisions at one point in time, often asking parents to reflect on decisions after the child's death, even though parents' understanding of prognosis and decisions about care evolve over time. We will evaluate parental decision-making for advanced cancer over time. 2) Existing work focuses on aggressive end-of-life care as the worst possible outcome. However, some parents wish to pursue aggressive measures even when they recognize that the child has little chance for cure. We will evaluate the extent to which parental decision-making for advanced cancer is informed and consonant with preferences, regardless of whether decisions lead to aggressive or palliative care. 3) Previous studies have focused on groups of different childhood cancers, making it difficult to ascertain whether differences in decision-making reflect differences in diseases, options for care, or parent preferences. We will focus on a single disease, relapsed neuroblastoma, as a model for parental decision-making. Children with relapsed neuroblastoma have advanced cancer but many options for care, including established cancer regimens, clinical trials, and palliation. Relapsed neuroblastoma presents an ideal model for parental decision-making in the setting of a complex array of choices. We will follow 120 parents at 8 institutions over time, beginning at relapse and continuing over 18 months. Parent interviews every 3 months and reviews of medical records throughout that time will be used to evaluate the ways that parental preferences for the aggressiveness of treatment change over time (Aim 1). Parental perception that care has been burdensome will be evaluated as possible driver of change in decision-making (Aim 2). Ideally, parent values for care would be the primary driver of treatment goals. Thus we will evaluate the extent to which parental understanding of prognosis, treatment options, and expected benefits and burdens of treatment can allow decision-making consonant with parental preferences in the absence of prior negative experiences with care (Aim 3). Finally, in-depth parent interviews will allow us to evaluate personal factors that drive parental decision-making (Aim 4). Throughout the study, a Parent Advisory Group will guide assessment of care preferences and decision-making.

ELIGIBILITY:
Inclusion Criteria:

* Parent of a child with relapsed or refractory high risk neuroblastoma, as defined by the International Neuroblastoma Risk Group, without respect to timing of first determination of relapse or refractory disease;
* Parent aged 18 years or older, of a child aged <=18 years;
* English- or Spanish-speaking.

Exclusion Criteria:

* Delirium/dementia as judged by the treating physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parents of children with relapsed or refractory neuroblastoma.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Number of parents who prefer life-prolonging care | 18 months
  Questionnaire-based measure

SECONDARY OUTCOMES:
Number of parents who experience decisional regret | 18 months
  Questionnaire-based measure
Number of parents who report that care has been burdensome | 18 months
  Questionnaire-based measure
Number of parents who report that care received is consonant with the parent's preferences | 18 months
  Questionnaire-based measure

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer W Mack, MD MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (9):
- United States (9):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Stanford/Packard's Children's Hospital, Palo Alto, California
  - The University of Chicago Medical Center, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Cook's Children's Healthcare System, Fort Worth, Texas
  - Seattle Children's Hospital, Seattle, Washington